CLINICAL TRIAL: NCT03026569
Title: Orange Juice as Dietary Source of Antioxidants for Patients With Hepatitis C Under Antiviral Therapy
Brief Title: Orange Juice Consumption in Patients With Hepatitis C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: São Paulo State University (Other)
Responsible Party: Principal Investigator, Thais Cesar, PhD, São Paulo State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SaoPSU11
Record Dates: First submitted 2017-01-17; First posted 2017-01-20 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Infection
Keywords: orange juice; chronic hepatitis C; biochemical markers; oxidative stress; nutritional status; antioxidants
MeSH Terms: conditions — Persistent Infection; Hepatitis C, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Orange juice (Experimental): Orange juice: twenty-three patients with chronic hepatitis C under pegylated interferon combined with ribavirin treatment were supplemented with 100% commercial pasteurized orange juice (500 mL/d) during 8 weeks.
  Interventions: Other: Orange juice (500 mL/d)
- Control (No Intervention): Control: twenty patients with chronic hepatitis C under pegylated interferon combined with ribavirin treatment were monitored for consumption of orange juice during 12 weeks.

INTERVENTIONS:
Other: Orange juice (500 mL/d) — The patients were instructed to drink orange juice in two daily portions during eight consecutive weeks. Patients from both groups were asked to maintain their usual lifestyle, diet, and physical activity, and they were checked weekly by the researcher's team. Assessments of anthropometric data, dietary intake, as well as blood sample collection for biochemical analysis were performed in all participants on the first and last day of the experiment.
  Arms: Orange juice

SUMMARY:
This study aimed to verify whether orange juice, source of citrus flavonoids and vitamin C, may contribute to the treatment of patients with chronic hepatitis C.

DETAILED DESCRIPTION:
Forty-three patients with chronic hepatitis C who were being treated with pegylated interferon combined with ribavirin, according to the Clinical Protocol and Therapeutic Guidelines for Viral Hepatitis C and Co-infections of the Brazilian Health Ministry were randomly divided into two parallel groups: (1) orange juice (n = 23), which were supplemented with orange juice (500 mL/d) for 8 weeks; (2) control group (n = 20) composed of patients that were not drinking orange juice regularly. The recruitment process began in February 2012, the intervention was carried out from May 2012 to July 2012, and the data analysis started in September 2012. The sample number took into account variances on total cholesterol with a type I error α = 0.05 and a type II error β = 0.2 (80% power) (Dourado et al., 2015). The minimum sample size should have 20 individuals per group (n = 40), considering an approximately 15% dropout rate. Primary and secondary endpoints were the reduction of total cholesterol and modification of biochemical markers, respectively. Kolmogorov Smirnov and Levene test assessed normality and homogeneity of data, respectively. Assessment of the data was performed in all participants on the first and last day of the experiment. All the parameters were compared between the juice group and the control group using General Linear Model of Repeated Measures Analysis. Differences in baseline patients' characteristics between the two groups were analyzed by One-way analysis of variance (ANOVA). The LSD signed rank post-test was used to assess significant changes in parameters after the start of treatment in each group, and the differences were considered statistically significant at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Detection of circulating HCV RNA
* Negative HBV surface antigen
* Negative antibodies to HIV

Exclusion Criteria:

* Co-infection with hepatitis B virus (HBV)
* Co-infection with hepatitis A virus (HAV)
* Co-infection with human immunodeficiency virus (HIV)
* Presence of diabetes mellitus,
* Presence of ascites
* Elevation in serum ferritin levels

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Total cholesterol | 8 weeks

SECONDARY OUTCOMES:
Body mass | 8 weeks
Body mass index | 8 weeks
% body fat | 8 weeks
Waist circumference | 8 weeks
Glucose | 8 weeks
Insulin | 8 weeks
HOMA-IR | 8 weeks
LDL-C | 8 weeks
HDL-C | 8 weeks
Triglycerides | 8 weeks
CRP | 8 weeks
alkaline phosphatase | 8 weeks
AST | 8 weeks
ALT | 8 weeks
gamma-GT | 8 weeks
TBARS | 8 weeks
ABTS | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thais B Cesar, Ph.D, Principal Investigator — Sao Paulo State University "Julio de Mesquita Filho"
Locations (1):
- Sao Paulo State University "Julio de Mesquita Filho", Araraquara, São Paulo, Brazil

REFERENCES:
- [Background] Dourado GK, Cesar TB. Investigation of cytokines, oxidative stress, metabolic, and inflammatory biomarkers after orange juice consumption by normal and overweight subjects. Food Nutr Res. 2015 Oct 20;59:28147. doi: 10.3402/fnr.v59.28147. eCollection 2015. PMID 26490535